CLINICAL TRIAL: NCT01116492
Title: Study of the Inflammatory Reaction in Standard vs Single Port Cholecystectomy for Uncomplicated Cholelithiasis
Acronym: Lap vs SILS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: G. Hatzikosta General Hospital (Other)
Responsible Party: Konstantinos Tsimogiannis MD, "G. Hatzikosta" General Hospital of Ioannina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: GH-1948-05
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Last update posted 2010-05-21 (Estimated); Status verified 2010-05

CONDITIONS: Cholelithiasis; Inflammatory Response
Keywords: SILS; Inflammatory reaction; a-defensins; SILS vs standard laparoscopic cholecystectomy
MeSH Terms: conditions — Cholelithiasis; Inflammation | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lap Group (Active Comparator): Patients in this group are operated for uncomplicated cholelithiasis with standard 4 port laparoscopic cholecystectomy
  Interventions: Other: Laparoscopic cholecystectomy
- SILS group (Active Comparator): Patients in this group are operated for uncomplicated cholelithiasis with Single Incision Laparoscopic Cholecystectomy
  Interventions: Other: Single incision laparoscopic cholecystectomy

INTERVENTIONS:
Other: Single incision laparoscopic cholecystectomy — One port placed through the umbilicus
  Arms: SILS group
Other: Laparoscopic cholecystectomy — Standard 4 port laparoscopic cholecystectomy
  Arms: Lap Group

SUMMARY:
This is a study of the inflammatory reaction in standard 4 port laparoscopic cholecystectomy vs Single Port Laparoscopic (SIL) cholecystectomy. It is assumed that the reduced trauma in SIL Cholecystectomy causes reduced inflammatory reaction compared to the 4 port laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Two groups of 20 patients each are included in this study. Pre operatively, 6 and 24 hours postoperatively, blood is taken from these patients, it is centrifuged and the plasma is taken. IL-6, a-defensins and CRP are measured for each sample.

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated cholelithiasis
* American Society of Anesthesiologists (ASA) I or II
* No previous operations in upper abdomen
* Body mass index (BMI) <30

Exclusion Criteria:

* Cholecystitis
* ASA > II
* BMI>30
* Previous operations in upper abdomen
* Previous operations in intestine

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- "G. Hatzikosta" General Hospital of Ioannina, Ioannina, Greece